CLINICAL TRIAL: NCT04656873
Title: Lineberger Comprehensive Cancer Center (LCCC) 1937: Immuno-Oncology Database and Bioregistry: Identifying Mechanisms of Autoimmune Diseases in the Era of Cancer Immunotherapy.
Brief Title: Immuno-Oncology Database and Bioregistry
Acronym: IOG
Status: Active, not recruiting | Type: Observational
Sponsor: UNC Lineberger Comprehensive Cancer Center (Other)
Collaborators: University of North Carolina, Chapel Hill (Other); North Carolina Translational and Clinical Sciences Institute (Other)
Responsible Party: Sponsor
Other Study IDs: LCCC1937; 18-0560 (Other: UNC Chapel Hill IRB)
Record Dates: First submitted 2020-11-18; First posted 2020-12-07 (Actual); Last update posted 2025-09-04 (Actual); Status verified 2025-08

CONDITIONS: Malignancy; Immune System Diseases; Autoimmune Diseases
Keywords: cancer; immunotherapy; immune checkpoint inhibitors; immune related adverse events; autoimmune diseases
MeSH Terms: conditions — Neoplasms; Immune System Diseases; Autoimmune Diseases | interventions — Surveys and Questionnaires

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 2 Years
Biospecimen Retention: Samples With DNA — cheek swab, blood, urine, feces, medical waste tissue/fluids, research biopsies.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- ICI treatment: Adult cancer patients starting ICI monotherapy or combination therapy at UNC Chapel Hill per clinical standard of care and willing to allow specimens from surplus tissue to be banked for research purposes (in the case of resections) AND willing to have additional specimens taken for research purposes (in the case of biopsies). Patients will be followed for samples and clinical data from medical records from before starting ICI therapy until 2 years after the end of ICI treatment.
  Interventions: Procedure: Biospecimen Collection; Other: Medical Chart Review; Other: Questionnaires/Surveys

INTERVENTIONS:
Procedure: Biospecimen Collection — Undergo collection of cheek swab, blood, urine, stool, and tissue samples for research
Other: Medical Chart Review — Periodic review of medical records for clinical parameters (labs, ICI dosing and frequency, occurrence, timing and type of irAE, irAE management, etc.) along with relevant demographic information (age, sex/gender, race/ethnicity, insurance type, etc.).
Other: Questionnaires/Surveys — Periodic self-report questionnaires/surveys for symptom tracking, quality of life, perinatal outcomes, etc.

SUMMARY:
Immunotherapy, especially immune checkpoint inhibitors (ICIs), are effective in treating many different types of cancers. ICIs fight cancer by driving the immune system into an "activated state" that makes it harder for tumor cells to hide and easier for the immune system to destroy them. In doing this, oncologists risk "over activation" where immune cells can cause side effects that could affect any part of the body. These are known as immune related adverse events (irAEs). While irAEs are a known risk of ICIs, scientists and doctors do not understand how they develop, who is more likely to get them, and what is the best way to manage them while still getting the anti-tumor effects from ICIs. The aim of this project is to build an infrastructure for researchers to collaborate in clinical, translational, and basic science research focused on understanding and managing immune related adverse events (irAEs). The investigators will collect research data and samples from patients who receive ICI treatment, including when patients might experience immunotherapy side effects, to store for use in future research studies.

DETAILED DESCRIPTION:
BACKGROUND

Tumors evolve to evade the body's anti-tumor immune response by targeting cancer cells and downregulating immune pathways. Immune checkpoint inhibitors (ICIs) prevent this tumor evasion by driving the immune system into an "activated state", and upregulating the patient's immune system to destroy tumor cells. While enhancing the immune system disrupts tumor growth, in doing so oncologists risk "over activation" resulting in immune-mediated toxicity known as immune related adverse events (irAEs).

irAEs are an emerging disease entity, affecting many organ systems with diverse clinical presentations similar to known autoimmune diseases, such as systemic lupus erythematosus, inflammatory arthritis, psoriasis, thyroiditis, inflammatory bowel disease, hepatitis, pneumonitis, and myocarditis. The most common presentations of irAEs are dermatologic (rashes), endocrine (hypo/hyper-active thyroid, hypophysitis, adrenal), and gastrointestinal (colitis). However, any organ system can be affected resulting in a wide array of irAEs.

Immunotherapy, especially ICIs, are being increasingly used in a wide variety of cancer therapy and have been found to effectively treat many different types of cancers. ICIs are monoclonal antibodies targeting cytotoxic T-cell lymphocyte antigen 4 (CTLA-4), programmed cell death protein 1 (PD-1) or programmed death ligand 1 (PD-L1) pathways. CTLA-4 and PD-1/PD-L1 are involved in deactivating T-cell and attenuating T-cell effector response, respectively. These are already being used to treat a wide range of cancers with several clinical trials currently underway examining response of additional cancer types to current ICIs as well as for developing new ICI treatments. The investigators anticipate that there will be additional immune checkpoint targets in the future given that some are already in clinical trials and the high interest in cancer immunotherapy.

The goal of this project is to collect, curate, and store data and specimens for future studies presented in separate protocols. This patient registry will provide biological specimens for biomarker analysis, immunophenotyping, genetic and microbiome analysis to understand development of autoimmune conditions. Clinical data can be used for epidemiological studies as well as clinical, functional, psychosocial and economic outcomes research regarding impact of ICIs and irAEs on cancer patients. Moreover, this infrastructure can inform the development of clinical algorithms and help determine the effectiveness of medical interventions targeting cancer outcomes and irAEs.

STUDY OUTLINE

Patients will be involved in the study from the time of consent (before starting ICI therapy) until 2 years after the end of ICI treatment. The investigators will collect clinical data (including demographic information, medical history, cancer diagnosis and treatment, management of adverse events, and outcomes), specimens (including blood, urine, stool, biofluids and/or tissue samples), and questionnaires at multiple time points. All patient data and samples will be linked by a de-identified study specific identifier (study ID) and will be stored indefinitely until used or patient withdraw from the study in writing.

STUDY OBJECTIVES

The overall goal of this project is to build an infrastructure that will provide resources for researchers at UNC Chapel Hill and beyond to conduct multidisciplinary clinical, translational, and basic research in elucidating pathways involved in cancer biology and irAEs.

ELIGIBILITY:
Inclusion Criteria:

* 18 years of age at time of enrollment
* Diagnosis of cancer
* Starting initial ICI therapy or re-starting ICI treatment after a 2-year gap (including off-label use) at UNC-CH using any currently FDA approved ICI's.

Exclusion Criteria:

* Prior ICI treatment within the last 2 years, including FDA approved ICIs and those under investigation (clinical trials).
* Known and untreated BSL-2+ communicable diseases (active/untreated latent TB, HIV, etc.) or other active infections.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Adult cancer patients starting ICI monotherapy or combination therapy at University of North Carolina at Chapel Hill (UNC-CH).
Sampling Method: Non-Probability Sample
Enrollment: 32 (Actual)
Dates: Start 2021-05-20 (Actual); Primary Completion 2026-06-04 (Estimated); Study Completion 2026-06-04 (Estimated)

PRIMARY OUTCOMES:
Number of Participants With Immune Checkpoint Inhibitor Treatment-Related Adverse Events as Assessed by CTCAE v5.0 | Up to 2 years after end of ICI treatment
  Clinical database with a linked specimen biorepository from this cohort - including management of irAEs and underlying cancer, irAE and cancer outcomes, surveys (PROs) and specimen collection from various time points during and after treatment.

CONTACTS AND LOCATIONS:
Overall Officials: Rumey C Ishizawar, MD, PhD, Principal Investigator — UNC Chapel Hill
Locations (1):
- Lineberger Comprehensive Cancer Center at University of North Carolina, Chapel Hill, Chapel Hill, North Carolina, United States

IPD SHARING:
Plan to Share IPD: Yes
Members of the UNC IOG will review and approve all proposals or similar justifying access to and use of data and/or specimens for ancillary projects and collaborations. Utilizing data or specimens will require a separate IRB application after approval by UNC IOG as well as any contracting necessary for data and material use.
  To start a request for use of research data and/or specimens, please complete form at the link below.
Supporting Information: Study Protocol, ICF
Time Frame: Upon request.
Access Criteria: Any pertinent regulatory agreements and approvals are in place.
URL: https://redcap.unc.edu/surveys/?s=4DCNA9J3WH

REFERENCES:
- See also: University of North Carolina Lineberger Comprehensive Cancer Center Clinical Trials — http://unclineberger.org/patientcare/clinical-trials/clinical-trials